CLINICAL TRIAL: NCT06914180
Title: Intravenous Infusion of Esketamine in Combination With Pulsed Radiofrequency for Trigeminal Postherpetic Neuralgia
Brief Title: Esketamine Combined With PRF for Trigeminal Postherpetic Neuralgia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Beijing Xiaotangshan Hospital (Other); The First Hospital of Fangshan District,Beijing (Other); Beijing Ditan Hospital (Other); Hengshui People's Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Day surgery and Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY-2024-332-02-03
Record Dates: First submitted 2025-03-25; First posted 2025-04-06 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Postherpetic; Neuralgia, Trigeminal (Etiology)
Keywords: trigeminal postherpetic neuralgia; esketamine
MeSH Terms: conditions — Neuralgia | interventions — Control Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esketamine group (Experimental): In addition to receiving PRF treatment+pregabalin, patients will also undergo a single intravenous infusion of esketamine
  Interventions: Drug: esketamine group
- control group (Placebo Comparator): patients will receive PRF treatment+pregabalin
  Interventions: Drug: control group

INTERVENTIONS:
Drug: esketamine group — In the esketamine group, in addition to receiving PRF treatment+pregabalin for rescue analgesia, patients will also undergo a single intravenous infusion of esketamine. A total of 0.5 mg/kg of esketamine will be diluted in 50 mL of normal saline. The infusion will commence with an intravenous injection of 10 mg of esketamine over 1 minute, followed by a maintenance dose of 8 mg/h. The infusion rate will be adjusted based on the patients' tolerance levels.
  Other Names: esketamine+PRF
  Arms: esketamine group
Drug: control group — In the control group, patients will receive PRF+pregabaline treatment. Pulsed radiofrequency (PRF) will be performed on GG by a designated physician in each participating center. PRF treatment (PMG-230, Baylis Medical Inc.) targeting to GG will be applied for 900 seconds. The parameters of PRF treatment will be set at 42 ℃, 2 Hz with 20 milliseconds current. Regarding pregabalin, the dosage is titrated based on patients'pain intensity and tolerance. This process fully accounts for individual patient differences to optimize treatment outcomes.
  Other Names: PRF
  Arms: control group

SUMMARY:
This trial's primary objective is to compare the analgesic efficacy of esketamine in combination with pulsed radiofrequency (PRF) against that of PRF monotherapy in patients with trigeminal postherpetic neuralgia (TPHN).

DETAILED DESCRIPTION:
This study aims to determine whether the addition of esketamine to the PRF regimen can relieve pain in TPHN patients. By doing so, the research endeavors to identify a rapid, effective, and safe treatment approach for refractory TPHN patients

ELIGIBILITY:
Inclusion Criteria:

1. Ages more than 18 years;
2. Pain persisting for over three months following the onset of the herpes zoster skin rash;
3. Lesions located in the trigeminal nerve or its branches innervated regions；
4. Having an average pain score of at least 4 on a Numeric Rating Scale (NRS, 0 = no pain, 10= worst possible pain)；
5. Planned to perform CT-guided PRF treatment of the gasserian ganglion(GG).

Exclusion Criteria:

1. Obstructive sleep apnoea syndrome;
2. Those who receive other more invasive treatments, such as radiofrequency thermocoagulation (RFT) of GG.
3. A history of systemic immune diseases, organ transplantation, or cancers;
4. A history of severe cardiopulmonary, hepatic, renal dysfunction or coagulation function disorder;
5. A history of schizophrenia, epilepsy, or myasthenia gravis, delirium;
6. Comorbid hyperthyroidism or phaeochromocytoma;
7. Recent history of drug abuse;
8. Having contraindications to esketamine;
9. Communication difficulties.
10. Women who are preparing for pregnancy, in the pregnancy or lactation period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
1.the difference between the means of the daily mean pain scores over the first 7 days, measured on an 11-point Numeric Rating Scale（NRS） | 7-day period
  NRS score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain

SECONDARY OUTCOMES:
average weekly NRS score | up to 12 weeks
  average weekly NRS score of each participants for rescue analgesia.NRS score is a way to quantify the degree of subjective feelings such as pain using numbers. Generally, 0 represents no pain, and 10 represents the most severe pain.A higher score indicates more severe pain
averaged weekly analgesic consumption | up to 12 weeks
  averaged weekly consumption per analgesic of each participant
the 12-item Short-Form Health Survey (SF-12) score | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  Quality of life (QoL) assessed by the SF-12 score(range 0-100, with higher scores indicating better health status)
the Pittsburgh Sleep Quality Index (PSQI) score | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  Sleep quality measured by PSQI score(range 0-21, with higher scores indicating poorer sleep quality)
the Patient Global Impression of Change scale (PGIC) | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  The Patient Global Impression of Change (PGIC) is usually a 7 - point scale. The scale title is "Patient Global Impression of Change". The minimum value is 1 and the maximum value is 7.In summary, for the PGIC scale, lower scores (from 1 to 3) mean a better outcome, indicating improvement in the patient's condition, while higher scores (from 5 to 7) mean a worse outcome, suggesting a deterioration of the condition. Score 4 represents a neutral state of no change.
the Hospital Anxiety and Depression Scale (HADS) | At the end of weeks 1, 2, 4, 8, and 12 after treatment
  It 6.consists of two sub-scales. Each sub-scale consists of 7 items and each item scored from 0 to 3. A higher score indicates more severe anxiety or depression. A score of 11 or above can indicate clinically significant anxiety or depression.
Safety assessments | Conducted on Day 0, Day 1, Day 3, and at the end of weeks 1, 2, 4, 8, and 12 after treatment
  intraoperative complications, PRF-related complications, Eskatamine-related complications, Pregabaline-related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not yet decided